CLINICAL TRIAL: NCT03054038
Title: Phase I Trial of Combination Afatinib and Necitumumab in EGFR Mutation Positive NSCLC With Acquired Resistance to First or Third Generation EGFR TKIs
Brief Title: Afatinib and Necitumumab in Patients With EGFR Mutation Positive Advanced or Metastatic Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Sally York, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 1684; NCI-2016-01532 (Other Grant/Funding Number: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2016-10-25; First posted 2017-02-15 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Non-Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; necitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patients receive afatinib PO QD on days 1-28 and necitumumab IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib; Biological: Necitumumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Afatinib — Given by mouth
Biological: Necitumumab — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of afatinib and necitumumab and to see how well they work in treating patients with EGFR mutation positive non-small cell lung cancer that has spread to other places in the body. Afatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as necitumumab, may interfere with the ability of tumor cells to grow and spread. Giving afatinib and necitumumab may work better in treating patients with EGFR mutation positive non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of combination afatinib and necitumumab therapy in EGFR mutation positive non-small cell lung cancer (NSCLC) patients who have progressed following first- and third-generation EGFR tyrosine kinase inhibitors (TKIs).

II. To determine the efficacy and safety profile of afatinib and necitumumab combination therapy in patients with EGFR mutation positive NSCLC patients who have progressed following first- and third-generation EGFR TKIs.

OUTLINE: This is a dose-escalation study.

Patients receive afatinib orally (PO) once daily (QD) on days 1-28 and necitumumab intravenously (IV) over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Histologically or cytologically-confirmed advanced or metastatic non-small cell lung cancer (NSCLC) that is EGFR mutation positive; rare sensitizing mutations allowed
* Progression on a first generation EGFR TKI (T790M negative), or progression on a third generation TKI (if T790M positive at time of progression on a first or second generation TKI)
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 that can be followed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Patient consents to undergo a medically safe tumor biopsy at time of disease progression for mutation analysis
* Leukocytes >= 3,000/uL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.5 g/dL
* Calculated creatinine clearance > 50 mL/min (per the Cockcroft-Gault formula)
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase (ALP) =< 3.0 x ULN
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3.0 x ULN; for patients with hepatic metastases, ALT and AST =< 5.0 x ULN are acceptable

  * Note: if a patient experiences elevated ALT > 5 x ULN and elevated total bilirubin > 2 x ULN, clinical and laboratory monitoring should be initiated by the investigator; for patients entering the study with ALT > 3 x ULN, monitoring should be triggered at ALT > 2 x baseline
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days prior to receiving first dose of study medication; and additionally agree to use at least two methods of birth control or abstain from heterosexual intercourse from the time of signing consent, and until 6 months after patient's last dose of study drug

  * WOCBP of childbearing potential are defined as those not surgically sterile or not post-menopausal (i.e. if a female patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for 24 months in the absence of an alternative medical cause, then patient will be considered a female of childbearing potential); postmenopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women
* WOCBP must agree to follow instructions for method(s) of contraception from the time of signing consent and until 6 months after last dose of study therapy
* Men able to father children who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception from the time of signing consent and until 6 months after last dose of study therapy; men able to father children are defined as those who are not surgically sterile (i.e. patient has not had a vasectomy)

Exclusion Criteria:

* Prior treatment against NSCLC with an EGFR monoclonal antibody
* Prior afatinib therapy, unless patient received an intervening third generation EGFR TKI after concluding prior afatinib and before enrollment on this clinical study
* Less than 3 days from prior treatment with EGFR TKI; patients with adverse events related to prior EGFR TKI must recover to Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 to be eligible
* History of arterial or venous thromboembolism within 3 months prior to study enrollment; patients with a history of venous thromboembolism beyond 3 months prior to study enrollment can be enrolled if they are appropriately treated with low molecular weight heparin
* Subjects with a history of interstitial lung disease (e.g., sarcoidosis) that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity; subjects with chronic obstructive pulmonary disease (COPD) whose disease is controlled at study entry are allowed
* Symptomatic brain metastases; stable and treated central nervous system (CNS) disease allowed; patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least two (2) weeks prior to initiating study treatment; anticonvulsant therapy will be allowed if patient is on a stable or decreasing dose of anticonvulsant treatment for at least two (2) weeks prior to initiating study treatment
* Subjects with carcinomatous meningitis
* Prior radiotherapy or radiosurgery < 2 weeks prior to starting study treatment
* Current symptomatic congestive heart failure (New York Heart Association classification >= grade III), unstable cardiac arrhythmia requiring therapy (e.g. medication or pacemaker), unstable angina (e.g. new, worsening or persistent chest discomfort), or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100 mmHg); or any of the following occurring within 6 months (180 days) prior to first dose of study treatment: myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack; use of antihypertensive medication to control blood pressure is allowed
* Patient is pregnant or breastfeeding, or plans to become pregnant or father children from time of signing consent and lasting until 6 months after the last dose of trial treatment
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured AND no additional therapy is ongoing and required during the study period with the exception of bisphosphonates and anti-androgens and/or gonadorelin analogues for the treatment of prostate cancer are permitted; subjects with other active malignancy requiring concurrent intervention are excluded
* Requiring treatment with any of the prohibited concomitant medications listed that cannot be stopped for the duration of trial participation
* Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhea, malabsorption)
* Recent (within 30 days before enrollment) or concurrent yellow fever vaccination
* All toxicities attributed to prior anti-cancer therapy other than alopecia, fatigue, or peripheral neuropathy must have resolved to grade 1 (National Cancer Institute [NCI] CTCAE version 4) or baseline before administration of study drug
* The patient has any ongoing or active infection, including active tuberculosis; Note: a urinary tract infection controlled with oral antibiotics initiated at least 7 days prior to study entry is acceptable
* Known positive test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)
* The patient has a known allergy/history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab, or any other contraindication to one of the administered treatments
* Known hypersensitivity to afatinib or the excipients of any of the trial drugs
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose experience a dose-limiting toxicity | Up to 28 days
  Highest dosage at which 0 or 1/6 patients

SECONDARY OUTCOMES:
Objective response rate | Up to one year
  Complete response assessed by RECIST version (v) 1.1
Objective response rate | Up to one year
  Partial response assessed by RECIST version (v) 1.1
Overall survival | From the first dose of study treatment to the time of death from any cause on study, assessed up to 1 year
  Assessed by RECIST v1.1
Duration of response | Up to 1 year
  Assessed by RECIST v1.1
Incidence of adverse events | Up to 1 year
  Assessed by NCI CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Sally York, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided